CLINICAL TRIAL: NCT03921229
Title: Feasibility, Acceptability, and Pilot Randomized Controlled Trial of a Tele-Coaching Intervention to Improve Treatment Adherence in Cystic Fibrosis
Brief Title: Tele-Coaching Intervention to Improve Treatment Adherence in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Johns Hopkins University (Other); University of Kansas Medical Center (Other); West Virginia University (Other)
Responsible Party: Principal Investigator, Gregory Sawicki, Co-Chair of Success with Therapies Research Consortium, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00031836; STRC-109-16-02 (Other: Success with Therapies Research Consortium)
Record Dates: First submitted 2019-04-04; First posted 2019-04-19 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
Keywords: Patient Care; Tele-health; Behavioral intervention
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 6-months of 11 web-based intervention (tele-coaching) sessions (9 biweekly sessions and 2 monthly sessions) of approximately 30 minutes each; continued use of eTrack nebulizer and vest monitor photo capture as measures of adherence.
  Interventions: Behavioral: Tele-coaching

INTERVENTIONS:
Behavioral: Tele-coaching — Patients will meet with a "tele-coach," who is a care team member, via video-calling, on a regular basis for six months to identify and address treatment adherence concern(s).

SUMMARY:
This is a prospective, multicenter pilot study to investigate the feasibility and preliminary effectiveness of a tailored tele-coaching intervention to enhance medical adherence in patients with CF.

DETAILED DESCRIPTION:
This is a prospective, multicenter pilot study to test the feasibility and acceptability of a tele-coaching intervention and its implementation in patients with CF (ages 14-25 years), and to obtain estimates of treatment effects across a range of key outcome measures (e.g., global adherence, change in treatment barriers, specific improvement in adherence, etc.)

ELIGIBILITY:
Inclusion Criteria:

COACH Participants:

1. Be a CF-focused clinician employed by one of the study sites, including: social workers; respiratory therapists, pharmacists, nurse practitioners, nurses, mental health coordinators, dieticians, and psychologists.

PATIENT Participants:

1. Male or female ≥ 14 and ≤ 25 years of age;
2. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria: (a) sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis test (QPIT), and/or (b) two well-characterized mutations in the CFTR (cystic fibrosis transmembrane conductance regulator) gene;
3. Has been prescribed one or more respiratory nebulized medications, such as: (a) dornase alfa, (b) hypertonic saline, (c) inhaled tobramycin, (d) inhaled aztreonam, (e) inhaled colistimethate *and/or* uses a vest device for airway clearance;
4. If taking, or anticipating to start on, Trikafta, has been taking the modulator for 6 weeks prior to enrolling in the study;
5. Has access to necessary resources for participating in a technology-based intervention: (a) mobile phone, tablet, computer, or digital camera capable of capturing and sending a digital image, and access to Internet; (b) an email account;
6. Is English-speaking;
7. Endorsed score of ≥3 on any treatment component on the CF-CBS at Enrollment Visit.

CAREGIVER Participants:

1. Is a caregiver of and resides with a Patient Participant in this study;
2. Has received permission from the Patient Participant, if aged 18 years of age or older, to be in the study; and
3. Is English-speaking.

Exclusion Criteria:

COACH Participants:

1. Anticipated change in CF Center during study period;
2. Physicians (MD, DO, or equivalent degree);
3. Advanced practice providers (e.g., APRN, PA) who serve as the primary provider in the CF clinic setting; and
4. Site research coordinator designated for this study.

PATIENT Participants:

1. Participation in the previous Tele-coaching study;
2. Anticipated transition to another CF care center within study period;
3. Planned or scheduled hospitalization between consent and start of intervention;
4. Self-reported current or planned pregnancy;
5. Having a person in the same household who is also enrolled in the study;
6. Presence of a condition, abnormality, or other factor that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data including, but not limited to: (a) diagnosis of intellectual or developmental disability that would preclude safe or adequate completion of measures; (b) history of, or planned, lung transplant;
7. Participation in concurrent studies targeting improvement in treatment adherence.

CAREGIVER Participants:

1. Participation in the previous Tele-coaching study;
2. Only one caregiver per Patient Participant can be enrolled in the Caregiver Cohort.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Patient attrition | up to 30 months
  Patient attrition will be measured as the percentage of participants who do not receive a sufficient dose of the intervention.
Intervention acceptability for patients assessed by Likert scale | up to 30 months
  This measure was developed for this specific study to evaluate feasibility and acceptability of the intervention through aspects of usability, quality, and satisfaction. Assessed by 5 point Likert Scale: Strongly disagree, Disagree, Neither Agree or Disagree, Agree, Strongly Agree.
Intervention acceptability for coaches assessed by Likert scale | up to 30 months
  This measure was developed for this specific study to evaluate feasibility and acceptability of the intervention through aspects of usability, quality, and satisfaction. Assessed by 5 point Likert Scale: Strongly disagree, Disagree, Neither Agree or Disagree, Agree, Strongly Agree.
Recruitment and feasibility | up to 30 months
  Recruitment and feasibility will be evaluated using the percentage of screen failures which are the number of eligible participants who do not score at least a three on any given treatment component for the CF-CBS amongst all eligible participants.

SECONDARY OUTCOMES:
Mean change in global adherence | Day 1 to approximately week 51
  Assess the preliminary effect of intervention on treatment adherence from data collected from vest photo capture and eTrack nebulizers. Vest photo capture will be scored as a ratio of total minutes used to total minutes prescribed in the study period. Medication adherence will be scored as a 'per drug analysis' of adherence with a ratio of competed to total prescribed doses in the study period. A composite score will be determined based on prescribed medications and medication/doses taken.
Change in treatment barriers | Day 1 to approximately week 51
  The CF-CBS (Cystic Fibrosis Care Behaviors Survey) will be used to analyze barriers to treatment. Measure will be based on an overall decrease (difference in means) in barrier specific frequency, specific treatment total barriers and the composite score for barriers from pre-intervention to post-intervention.

OTHER OUTCOMES:
Exploratory outcome: self-reported adherence | Day 1 to approximately week 51
  We will compare the Self-Reported Adherence measure and the CF-CBS Self-Reported Adherence using Pearson Correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Polineni, MD, MPH, Principal Investigator — University of Kansas Medical Center; Christina Duncan, PhD, Principal Investigator — West Virginia University
Locations (6):
- United States (6):
  - Stanford University, Palo Alto, California
  - National Jewish Health, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No